CLINICAL TRIAL: NCT06857916
Title: Cycling Intervention With Biofeedback of Power Symmetry for Patients With Stroke in an Inpatient Rehabilitation Facility: Pilot Randomized Controlled Trial.
Brief Title: Cycle and Stroke With Biofeedback for Power Symmetry
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00135445
Record Dates: First submitted 2022-12-28; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Stroke
Keywords: cycling; power; inpatient rehabilitation; biofeedback; gait symmetry
MeSH Terms: conditions — Stroke | interventions — Biofeedback, Psychology

STUDY DESIGN:
Intervention Model Description: pilot randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional rehabilitation (Active Comparator): Participants will undergo traditional rehabilitation therapies in the inpatient rehabilitation facility.
  Interventions: Other: Traditional
- cycle with biofeedback (Experimental): Participants will undergo traditional rehabilitation therapies in the inpatient rehabilitation facility. They will also participate in the cycle intervention with biofeedback. This will take place as an additional rehabilitation session.
  Interventions: Other: cycle with biofeedback

INTERVENTIONS:
Other: Traditional — Traditional rehabilitation course will occur.
  Arms: Traditional rehabilitation
Other: cycle with biofeedback — Individuals will receive biofeedback about their power production and power symmetry while participating in a 32 minute recumbent cycling session in inpatient rehabilitation facility.
  Arms: cycle with biofeedback

SUMMARY:
To determine changes in power symmetry, gait symmetry, and functional outcomes for participants' poststroke (Inpatient Rehabilitation Facility) after participating in an intervention using a recumbent cycle with power biofeedback (BFB). To determine how this intervention can impact gait asymmetry, a common disorder poststroke secondary to hemiparesis. Gait asymmetry is a difficult impairment to treat because it is difficult for both therapists and patients to perceive. Training with BFB allows for quantitative data about the power production or lack of that directly impacts safety in walking, increased energy expenditure, and decreased gait speed.

DETAILED DESCRIPTION:
Specific Aim 1 will determine the change in cycling power using BFB on a group of participants with stroke in an Inpatient Rehabilitation Facility. Specific Aim 2 will determine the effect size of the change in gait symmetry with cycling training with power BFB pre- to post-cycle intervention. Specific Aim 3 will determine the effect size of the change in functional mobility with cycling training with power BFB pre- to post-cycle intervention. Understanding the impact of cycle training with power BFB is an important step in improving stroke rehabilitation. This study is significant because it will provide data about power asymmetries in participants' early post-acute stroke and the transfer of training with power BFB to gait impairments.

ELIGIBILITY:
Inclusion Criteria:

1. they have a confirmed MCA or ACA ischemic or intracerebral hemorrhagic stroke, confirmed by CT/MRI or clinical documentation

   -AND demonstrating lower extremity hemiparesis [< 100 on lower limb Motricity Index24]
2. 18 to 70 years of age
3. a Functional Ambulation Category of 2 (Dependent Level II) through 5 (Independent Level surfaces only)
4. medical clearance to participate

Exclusion Criteria:

1. contractures that limit lower limb range of motion
2. cardiovascular, respiratory or metabolic instability, including unstable angina or hypertension above 200/110 at rest
3. uncontrolled diabetes
4. severe respiratory disorders that limit exercise
5. inability to ambulate > 150 feet prior to stroke
6. prior history of peripheral or central nervous system injury
7. moderate to severe hemispatial neglect according to the Kessler Foundation Neglect Assessment
8. major cognitive impairment preventing the capability to understand training instructions; identified by inability to follow 3-step command
9. severe aphasia preventing communication with the therapist.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-11-14 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in cycling power | pre- (admission day 2) and post- (day 14)
  Determine the change in cycling power using Biofeedback (BFB) on a group of participants with stroke in an Inpatient Rehabilitation Facility
Change in gait symmetry | pre- (admission day 2) and post- (day 14)
  Determine the effect size of the change in gait symmetry pre- to post-intervention after cycling with Biofeedback (BFB). Participants will be assessed on gait symmetry patterns (magnitude and timing of propulsion), using an instrumented treadmill (Bertec).

CONTACTS AND LOCATIONS:
Overall Officials: Heather A Hayes, PhD, Principal Investigator — University of Utah; James C Martin, PhD, Principal Investigator — University of Utah
Locations (1):
- University Health, Neilsen Rehabilitation Hospital, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No